CLINICAL TRIAL: NCT00826943
Title: Is Levocetirizine Less Sedating Than Cetirizine? A Randomized, Double-blind, Placebo Controlled Trial.
Brief Title: Is Levocetirizine Less Sedating Than Cetirizine?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Douglas Tzanetos, Fellow, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 080829
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Cetirizine; levocetirizine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Levocetirzine (Active Comparator): 5 mg daily x 7 days (note = cross over = all participants receive active comparators and placebo)
  Interventions: Drug: Levocetirizine
- cetirizine (Active Comparator): 10 mg daily x 7 days. Note = crossover study, so all participants recieve all active comparators and placebo.
  Interventions: Drug: Cetirizine
- placebo (Placebo Comparator): one tablet daily x 7 days; note that this is a crossover study so all participants receive all active comparators and placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cetirizine — Cetirizine 10 mg tab daily x 7 days
  Arms: cetirizine
Drug: Levocetirizine — 5 mg tab daily x 7 days
  Arms: Levocetirzine
Drug: Placebo — Placebo tablet daily x 7 days
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether cetirizine (zyrtec), levocetirizine (xyzal), and placebo differ in the degree of sedation they produce and their relief of allergy symptoms.

DETAILED DESCRIPTION:
Levocetirizine, the R-enantiomer of cetirizine, has been found to be less sedating relative to placebo than was cetirizine in separate trials. We plan to examine whether patients who did not tolerate cetirizine due to sedation are able to tolerate levocetirizine. This study will utilize a randomized, double-blind, placebo controlled trial comparing levocetirizine, cetirizine, and placebo in regards to sedation and allergy symptom scores. Each patient will receive levocetirizine, cetirizine, and placebo in randomized order and thus serve as their own control.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years of age or older
* patients with perennial allergic rhinitis sensitized (positive RAST within the last 3 years or wheal greater than or equal to 3 mm within the last 3 years) to either:

  * dust mite
  * cat (if they own an indoor cat)
  * dog (if they own an indoor dog)
* will allow for sensitization to tree, grass, or weed pollen, cockroach, or mold
* history of reported sedation/somnolence when taking cetirizine
* patient must have taken cetirizine for at least 1 week prior to discontinuing it
* patients must have either tolerated levocetirizine in the past or have never tried levocetirizine.

Exclusion Criteria:

* chronic urticaria requiring ongoing antihistamine or steroid treatment
* atopic dermatitis requiring ongoing antihistamine or steroid treatment
* URI or sinus infection during the 2 weeks preceding the beginning of the study
* vasomotor (non-allergic) or irritant rhinitis
* afrin use
* elderly or over 77 years of age (could affect creatinine clearance) or chronic renal insufficiency
* patients who have not tolerated levocetirizine in the past due to sedation.
* taking other prescription or over the counter antihistamines and unwilling to stop them during the study
* the presence of a sleep disorder such as sleep apnea or narcolepsy
* the use of as needed sleeping aid medication
* the presence of other chronic medical conditions which in the opinion of the investigator would prevent the subject from being able to participate effectively

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas B Tzanetos, M.D., Principal Investigator — Vanderbilt University Medical Center; John M Fahrenholz, M.D., Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Asthma, Sinus, and Allergy Clinic, Nashville, Tennessee, United States

REFERENCES:
- [Background] Devalia JL, De Vos C, Hanotte F, Baltes E. A randomized, double-blind, crossover comparison among cetirizine, levocetirizine, and ucb 28557 on histamine-induced cutaneous responses in healthy adult volunteers. Allergy. 2001 Jan;56(1):50-7. doi: 10.1034/j.1398-9995.2001.00726.x. PMID 11167352
- [Background] de Blic J, Wahn U, Billard E, Alt R, Pujazon MC. Levocetirizine in children: evidenced efficacy and safety in a 6-week randomized seasonal allergic rhinitis trial. Pediatr Allergy Immunol. 2005 May;16(3):267-75. doi: 10.1111/j.1399-3038.2005.00216.x. PMID 15853959
- [Background] Bachert C, Bousquet J, Canonica GW, Durham SR, Klimek L, Mullol J, Van Cauwenberge PB, Van Hammee G; XPERT Study Group. Levocetirizine improves quality of life and reduces costs in long-term management of persistent allergic rhinitis. J Allergy Clin Immunol. 2004 Oct;114(4):838-44. doi: 10.1016/j.jaci.2004.05.070. PMID 15480324

RESULTS

PARTICIPANT FLOW:
Groups:
- L Then C Then P: Levocetirizine 5 mg daily x 7 days then cetirizine 10 mg daily x 7 days then placebo daily x 7 days (wash out periods before and after each)
- L Then P Then C: Levocetirizine 5 mg daily x 7 days then placebo daily x 7 days then cetiriznie 10 mg daily x 7 days (wash out periods before and after each)
- P Then L Then C: placebo daily x 7 days then levocetirizine 5 mg daily x 7 days then cetirizine 10 mg daily x 7 days (wash out periods before and after each)
- P Then C Then L: placebo daily x 7 days then cetirizine 10 mg daily x 7 days then levocetirizine daily x 7 days (wash out periods before and after each)
- C Then L Then P: cetirizine 10 mg daily x 7 days then levocetirizine 5 mg daily x 7 days then placebo daily x 7 days (wash out periods before and after each)
- C Then P Then L: cetirizine 10 mg daily x 7 days then placebo daily x 7 days then levocetirizine 5 mg daily x 7 days (wash out periods before and after each)
Period: Overall Study
Arm/Group | L Then C Then P | L Then P Then C | P Then L Then C | P Then C Then L | C Then L Then P | C Then P Then L
Started | 6 | 6 | 4 | 5 | 7 | 2
Completed | 6 | 6 | 4 | 5 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Cross Over (all participants received all interventions)
Arm/Group | All Study Participants
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Secondary Outcome: Total Four Symptom Scores (Allergy Symptoms)
Description: Total Four Symptom Scores (TFSS) ranging 0 to 12. Increased scores indicate increased symptoms. This was measured on days 5, 12, 17, 24, 29, and 36 of the study. The mean TFSS for patients receiving placebo, cetirizine, and levocetirizine was then calculated.
  This was mean data for all interventions.
Time Frame: same as primary outcome measure (obtain on days 5, 12, 17, 24, 29, and 36)
Measure: Mean (Standard Deviation); unit: TFSS scores
Groups:
- Placebo; Levocetirizine: Cross Over (all participants received all interventions)
- Cetirizine: cross over = all participants received all interventions
Arm/Group | Placebo | Levocetirizine | Cetirizine
Number analyzed (Participants) | 29 | 29 | 29
TFSS scores | 4.41 (3.76) | 3.14 (2.67) | 2.67 (2.44)
Statistical Analysis 1: Comparison: Placebo vs Cetirizine; Test type: Superiority or Other; p = .03, Wilcoxon (Mann-Whitney) — The threshold for significance was p < 0.05
Statistical Analysis 2: Comparison: Placebo vs Levocetirizine; Test type: Superiority or Other; p = .11, Wilcoxon (Mann-Whitney) — The threshold for significance was p < 0.05
Statistical Analysis 3: Comparison: Levocetirizine vs Cetirizine; Test type: Superiority or Other; p = .45, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Modified Epworth Sleepiness Scale
Description: Epworth Sleepiness Scale ratings (0 to 24); higher scores = increased sedation. This was measured over the 36 days of the study (at the end of each washout period and each intervention period); measured on days 5, 12, 17, 24, 29, and 36.
  This was mean data for all interventions.
Time Frame: 36 days of the study
Population: per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Levocetirizine | Cetirizine
Number analyzed (Participants) | 29 | 29 | 29
units on a scale | 6.14 (4.58) | 6.69 (4.05) | 7.48 (5.31)
Statistical Analysis 1: Comparison: Placebo vs Cetirizine; Test type: Superiority or Other; p = .27, Wilcoxon (Mann-Whitney) — The threshold for significance was p < .05
Statistical Analysis 2: Comparison: Placebo vs Levocetirizine; Test type: Superiority or Other; p = .8, Wilcoxon (Mann-Whitney) — The threshold for significance was p < 0.05
Statistical Analysis 3: Comparison: Levocetirizine vs Cetirizine; Test type: Superiority or Other; p = .52, Wilcoxon (Mann-Whitney) — The threshold for significance was p < 0.05

3. Primary Outcome: Likert Score Rating Global Sedation
Description: Likert score range 1 to 9 (no sedation to extreme sedation). Highers scores indicate increased sedation. This was measured on days days 5, 12, 17, 24, 29, and 36 of the study.
  This was mean data for all interventions.
Time Frame: duration of study (36 days)
Population: per protocol
Measure: Mean (Standard Deviation); unit: Likert score
Arm/Group | Placebo | Levocetirizine | Cetirizine
Number analyzed (Participants) | 29 | 29 | 29
Likert score | 2.80 (1.67) | 3.07 (1.92) | 3.54 (2.17)
Statistical Analysis 1: Comparison: Placebo vs Cetirizine; Test type: Superiority or Other; p = .14, Wilcoxon (Mann-Whitney) — The threshold for significance was p < 0.05
Statistical Analysis 2: Comparison: Placebo vs Levocetirizine; Test type: Superiority or Other; p = .54, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Levocetirizine vs Cetirizine; Test type: Superiority or Other; p = .42, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Placebo | Levocetirizine | Cetirizine
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No